CLINICAL TRIAL: NCT05781893
Title: BALCoS - Basel Long COVID Cohort Study and DiLCoS - Digital Long COVID Substudy
Brief Title: Basel Long COVID-19 Cohort Study and Digital Long COVID Substudy
Acronym: BALCoS/DiLCoS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: State Secretariat for Education Research and Innovation, Switzerland (Other); European Union's Horizon Europe research and innovation programme (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2023-00359; th22Schaefert
Record Dates: First submitted 2023-03-20; First posted 2023-03-23 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Post COVID-19 Condition (PCC)
Keywords: Coronavirus disease (COVID); Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2); Somatic Symptom Disorder (SSD); fatigue; shortness of breath; cognitive dysfunction
MeSH Terms: conditions — Fatigue; Dyspnea; Cognitive Dysfunction | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for further analyses: genome and HLA typing (plasma), COVID-19 antibody profiling (serum), lipidome (serum), autoantibody epitopes (serum), and citrated plasma for coagulation analyses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BALCoS w/o DiLCoS: Patients of the cohort that are not enrolled in the DiLCoS substudy
  Interventions: Other: Data collection
- BALCoS w/ DiLCoS: Patients of the cohort that are additionnaly enrolled in the DiLCoS substudy
  Interventions: Other: Digital intervention (DiLCoS); Other: Data collection

INTERVENTIONS:
Other: Digital intervention (DiLCoS) — The DiLCoS substudy comprises a digital intervention. A smartphone app is used to provide the patient with a 12-week exercise program, including physical elements (in the form of breathing exercises, relief positions and relaxation techniques), psychoeducational elements (e.g., information about fatigue, neurocognitive symptoms, media consumption, healthy diet), self-monitoring elements (activity planning, energy management), and psychological elements (e.g., guided exercises to improve acceptance of current situation, cognitive distancing from negative thoughts, imagination techniques for pain management). It holds promise for significantly improving the management and quality of life of individuals living with PCC.
  Groups: BALCoS w/ DiLCoS
Other: Data collection — Data collection on sociodemography, clinical data (retrieved from regular care for PCC in the UHB medical outpatient clinic), biomarkers derived from blood samples, neurocognitive testing, psychometric questionnaires, and measures of physical performance.

SUMMARY:
The Basel Long COVID Cohort Study (BALCoS) is a registry-based cohort study that focuses on the patients' present health status, symptoms, the course of these symptoms, and potential mechanisms involved. The project aims to investigate proposed mechanisms behind Post COVID-19 condition (PCC), including a) autoimmunity, b) chronic inflammation, c) genetics, d) coagulation disorders, and e) psychosocial factors. Patients in the cohort can also join the Digital Long COVID Study (DiLCoS), a single-arm, cohort-based proof-of-feasibility study that is part of the larger BALCoS. DiLCoS is a intervention substudy designed to evaluate whether doing exercises delivered via a smartphone app (referred as digital intervention) can help with PCC. The digital intervention is a 12-week program that includes different kinds of exercises like breathing exercises, relaxation techniques, and tips on managing fatigue and other symptoms. It also teaches patients how to monitor their activities and energy levels, and provides psychological exercises to cope with negative thoughts and pain. Patients in the cohort complete a set of assessments that include the collection of sociodemographic and clinical data, biomarkers, neurocognitive testing, psychometric questionnaires, and measures of physical performance, and provide consent that their data from routine clinical care can be used for the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with PCC will be included. PCC will be defined as:
* History of confirmed or suspected SARS CoV-2 infection
* Symptoms usually start within 3 months from the onset of acute SARS CoV-2 infection with symptoms and effects that last for at least 2 months
* Symptoms cannot be explained by an alternative diagnosis
* signed informed consent is required

Additional Inclusion Criteria for participtation in DiLCoS:

* A smartphone with a compartible-operating system
* Separate signed informed consent is required

Exclusion Criteria:

* Age <18 years
* Lack of consent to participate in the study
* Language barriers (lack of sufficient knowledge of German)
* Lack of general understanding of study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited at the medical outpatient clinic unit at the UHB from April 2023 on. Any patient fulfilling inclusion criteria and lacking exclusion criteria will be asked to participate in the study and the substudy.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-04-20 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change in World Health Organization Disability Assessment Schedule (WHODAS 2.0) (12- item version) | At Baseline, T1 (BL + 3 months), T2 (BL + 6 months); T3 (BL + 12 months)
  The World Health Organization Disability Assessment Schedule (WHODAS 2.0) assesses and classifies disability due to health problems during the past 4 weeks. This study will utilize the 12- item version. Items are answered on a 5-point scale ranging from 0 = "none" to 4 = "extreme or cannot do".

OTHER OUTCOMES:
Change in Visual analogue scales (VAS) | At Baseline, T1 (BL + 3 months), T2 (BL + 6 months); T3 (BL + 12 months)
  Patients will answer 4 questions on a VAS with a rating slider ranging from 0 to 10. The questions will inquire symptom intensity (10 = it can't be worse), functional impairment (10 = can't be worse), quality of life (10 = can't be better), and work capacity (10 = full work capacity).
Change in EuroHIS Quality-of-Life-8 (QOL-8) | At Baseline, T1 (BL + 3 months), T2 (BL + 6 months); T3 (BL + 12 months)
  This 8-item instrument assesses quality of life and perceived health during the past 4 weeks. Items are answered on a 5-point scale, with wording differing between questions (e.g., from "very dissatisfied" to "very satisfied").
Change in the Somatic Symptom Disorder Questionnaire (SSD-12) | At Baseline, T1 (BL + 3 months), T2 (BL + 6 months); T3 (BL + 12 months)
  SSD-12 assesses psychological features of somatic disorders, e.g. catastrophizing thoughts and health anxiety. Items are answered on a 5-point scale ranging from 0 = "never" to 4 = "very often".
Change in the Patient Health Questionnaire (PHQ-15) | At Baseline, T1 (BL + 3 months), T2 (BL + 6 months); T3 (BL + 12 months)
  PHQ-15 assesses somatic symptom severity during the past 4 weeks. Patients are asked how impaired they felt by their symptoms, e.g. back pain. Items are answered on a 3-point scale ranging from 0 = "not bothered at all" to 2 = "bothered a lot".
Change in the Patient Health Questionnaire Depression Scale (PHQ-8) | At Baseline, T1 (BL + 3 months), T2 (BL + 6 months); T3 (BL + 12 months)
  PHQ-8 assesses the severity of depressive disorders. Patients are asked if in the past weeks, they were bothered by a problem. Items are answered on a 4-point scale ranging from 0 = "not at all" to 3 = "nearly every day".
Change in the Generalized Anxiety Disorder Questionnaire (GAD-7) | At Baseline, T1 (BL + 3 months), T2 (BL + 6 months); T3 (BL + 12 months)
  GAD-7 assesses if the patient was bothered by complaints related to anxiety during the past 2 weeks. Items are answered on a 4-point Likert scale ranging from 0 = "not at all" to 3 = "nearly every day".
Change in the Resilience Scale (Resilience Scale (RS-11) | At Baseline, T1 (BL + 3 months), T2 (BL + 6 months); T3 (BL + 12 months)
  The 11-item RS-11 asks about general resilience towards life events. Items are answered on a 7-point scale ranging from 1 = "strongly agree" to 7 = "strongly disagree".
Change in the Insomnia Severity Index (ISI) | At Baseline, T1 (BL + 3 months), T2 (BL + 6 months); T3 (BL + 12 months)
  Insomnia, e.g. difficulty falling asleep, is assessed by the ISI. Items are answered on a 5-point scale with regards to severity during the past 2 weeks, with wording differing between questions (e.g., from 0 = "very dissatisfied" to 4 = "very satisfied").
Change in the Chalder Fatigue Scale | At Baseline, T1 (BL + 3 months), T2 (BL + 6 months); T3 (BL + 12 months)
  Fatigue is assessed by the 11-item Chalder Fatigue Scale. Items are answered on a 4-point scale ranging from 0 = "Better than usual" to 3 = "much worse than usual".
Change in the Perceived Stress Scale (PSS) | At Baseline, T1 (BL + 3 months), T2 (BL + 6 months); T3 (BL + 12 months)
  The PSS investigates the experience of psychological stress in the past 4 weeks. It consists of 10 items. Items are answered on a 5-point scale ranging from 1 = "never" to 5 = "very often".
Change in JAMAR® grip strength test on the dominant hand | At Baseline and T3 (BL + 12 months)
  Grip strength will be assessed using the JAMAR®, a hydraulic grip strength measuring device (American Society for Surgery of the Hand, 1983). The test is repeated thrice for the dominant hand. The best value (in kg) is taken.
Change in 6-minute walking test | At Baseline and T3 (BL + 12 months)
  6-minute walking test is to assess functional exercise capacity by measuring the distance (in meters total) that a patient can walk in 6 minutes. Well-being before and after the test is assessed on a 5-point Likert-scale ranging from 1 = "very bad" to 5 = "very good". After the test, perceived exertion of breathing and legs is assessed with the Borg Category-Ratio (CR) 10 Scale ranging from 0 = "no exertion" to 10 = "maximal exertion"
Change in one minute sit-to-stand test (STS-60) | At Baseline and T3 (BL + 12 months)
  STS-60 is a measure for muscular endurance. It assesses the number of sit-to-stand cycles that can be achieved within one minute.
Change in neurocognitive status of patients assessed by CNS Vital Signs (CNSVS) test | At Baseline and T3 (BL + 12 months); approximately 40-50 minutes per test battery
  CNSVS is a computerized neurocognitive test battery that was developed as a routine clinical screening instrument. It consists of seven scientifically valid and reliable neuropsychological tests that normally require an interviewer. The tests are:
  verbal and visual memory, finger tapping, symbol digit coding, the Stroop Test, a test of shifting attention, and the continuous performance test. The Neurocognition Index reflects the overall or global neurocognitive functioning of the test taker. It is an average or the standard scores for five of the domains (composite memory, psychomotor speed, reaction time, complex attention and cognitive flexibility) that reflect the patient's performance on each assessment. CNS Vital Signs standardized have a mean of 100 and a standard deviation is 15. Higher scores are always better.
(Only BALCoS w/ DiLCoS) Progress and patients' engagement assessed by weekly feedback questions | After BL and before T1; at day 6 in weeks 1-11
  Patients enrolled in DiLCoS are presented with questions for qualitative feedback at the end of each weekly module within the digital intervention

CONTACTS AND LOCATIONS:
Overall Officials: Gunther Meinlschmidt, Principal Investigator — University Hospital Basel, Department of Psychosomatic Medicine
Locations (1):
- University Hospital Basel, Department of Psychosomatic Medicine, Basel, Switzerland

REFERENCES:
- [Derived] Rohner S, Schnepper R, Meinlschmidt G, Schaefert R, Mayr M, Bopp K, Meienberg A. Basel Long COVID Cohort Study (BALCoS): protocol of a prospective cohort study. BMJ Open. 2025 Jul 10;15(7):e093981. doi: 10.1136/bmjopen-2024-093981. PMID 40645616